CLINICAL TRIAL: NCT03192514
Title: Electronic Deprescribing Tool for the Prevention of Potentially Inappropriate Prescribing for Older Patients: A Protocol for a Cluster Randomized Trial
Brief Title: Electronic Deprescribing Tool for the Prevention of PIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting of family doctors below our goal
Sponsor: University of Beira Interior (Other)
Responsible Party: Principal Investigator, Luís Miguel André Monteiro, PhD Candidate at University of Beira Interior; Family Doctor, University of Beira Interior
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 31/17
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Prevention; Benzodiazepine Dependence
Keywords: Polypharmacy; Benzodiazepine use

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic Deprescribing tool (Experimental): GPs of enrolled patients with access to the electronic Deprescribing tool
  Interventions: Other: Electronic Deprescribing tool
- Usual Care (No Intervention): Usual care By GP´s

INTERVENTIONS:
Other: Electronic Deprescribing tool — Each GP of the intervention group will have exclusive access to an electronic tool that will guide them on deprescribing. The innovative electronic tool created by the researchers provide the rationale on indications for prescribing or deprescribing Benzodiazepines or/and Non-benzodiazepine hypnotics and also provides an interactive tapering suggestion integrated on a calendar.
  The tool emphasizes that any decision to continue or discontinue a drug remains a shared decision between GP and the patient.
  The electronic Deprescribing tool is designed to support clinical decisions
  Arms: Electronic Deprescribing tool

SUMMARY:
This study is a cluster randomized control trial aimed to measure the effectiveness of an educational knowledge transfer intervention to prescribers on the discontinuation of two targeted classes: Benzodiazepines andNon-benzodiazepine hypnotics.

DETAILED DESCRIPTION:
The investigators intend to develop an electronic decision support tool based on the best evidence available. This electronic deprescribing tool provides the rationale on the indications of prescribing or deprescribing Benzodiazepines or/and Non-benzodiazepine hypnotics and also provides interactive tapering suggestion integrated on a calendar. It is designed to help family doctors with the goal of improving health outcomes for the elderly.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥65 years who have been taking Benzodiazepines or/and Non-benzodiazepine hypnotics for at least 3 months and who do not meet any exclusion criterion

Exclusion Criteria:

* incapacity or unwillingness to provide written informed consent. Patient with dementia, psychotic disorder, a severe personality disorder; institutionalization; terminal illness, seizure disorders, rapid eye movement sleep disorders, benzodiazepine withdrawal, ethanol withdrawal, severe generalized anxiety disorder, epilepsy and periprocedural anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of benzodiazepine and Non-benzodiazepine hypnotics consumption at 3 months | 3 months
  The effectiveness of a new deprescribing electronic knowledge transfer tool for GP´s (rate of benzodiazepine and Non-benzodiazepine hypnotics discontinuation
Change from baseline of benzodiazepine and Non-benzodiazepine hypnotics consumption at 6 months | 6 months
  The effectiveness of a new deprescribing electronic knowledge transfer tool for GP´s (rate of benzodiazepine and Non-benzodiazepine hypnotics discontinuation
Change from baseline of benzodiazepine and Non-benzodiazepine hypnotics consumption at 12 months | 12 Months
  The effectiveness of a new deprescribing electronic knowledge transfer tool for GP´s (rate of benzodiazepine and Non-benzodiazepine hypnotics discontinuation

SECONDARY OUTCOMES:
Health-related quality of life of patients | At baseline, 3 months, 6 months, 12 months
  EQ-5D is a self-report questionnaire for measuring health-related quality of life
number of falls of patients | At baseline, 3 months, 6 months, 12 months
  Number of falls
motor vehicle crashes of patients | At baseline, 3 months, 6 months, 12 months
  Accidents recorded
Adverse drug withdrawal effects | At baseline, 3 months, 6 months, 12 months
  Any clinical effect
GPs level satisfaction regarding deprescribing | At baseline, 12 months
  Questionnaire with multiple choice, and open text format questions
Patients Beliefs about Medicines | At baseline, 3 months, 6 months, 12 months
  Beliefs about Medicines Questionnaire (BMQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Luís Monteiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No